CLINICAL TRIAL: NCT00704301
Title: Rivastigmine for Delirium in Intensive Care Patients, a Double-blind, Randomized Placebo-controlled add-on Trial
Brief Title: Rivastigmine for Intensive Care Unit (ICU) Delirium
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study is prematurely terminated due to a safety issue
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Novartis (Industry); Netherlands Brain Foundation (Other)
Responsible Party: Dr. A.J.C. Slooter, university Medical Center Utrecht, the Netherlands
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IC-DEL/009
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2009-10

CONDITIONS: Delirium
Keywords: Delirium; Confusion
MeSH Terms: conditions — Delirium; Confusion | interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Haloperidol: aged 70 years or less: 1 mg haloperidol three times a day i.v. older than 70 years: 0,5 mg haloperidol three times a day i.v. Rivastigmine: two times 1,5 mg a day; The dosage will be increased every three days with 3 mg a day, until the CAM-ICU is negative or until the occurrence of presumed severe adverse effects or until a maximum of 12 mg a day.
  Interventions: Drug: Rivastigmine
- 2 (Placebo Comparator): Haloperidol: aged 70 years or less: 1 mg haloperidol three times a day i.v. older than 70 years: 0,5 mg haloperidol three times a day i.v. Placebo: 2 times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivastigmine — Rivastigmine, two times 1,5 mg a day. The dosage will be increased every three days with 3 mg a day, until the CAM-ICU is negative or until the occurrence of presumed severe adverse effects or until a maximum of 12 mg a day.
  Other Names: Exelon
  Arms: 1
Drug: Placebo — Placebo, 2 times a day
  Arms: 2

SUMMARY:
Delirium in Intensive Care (IC) patients is a frequent disorder. The aim of this study is to investigate whether treatment of delirium in the ICU with rivastigmine added to haloperidol shortens the duration of delirium in comparison to placebo added to the treatment with haloperidol.

DETAILED DESCRIPTION:
Objective: To study whether rivastigmine added to treatment with haloperidol shortens the duration of delirium in ICU patients and reduces costs.

Study design: Multicentre, double-blind, randomized controlled trial. Study population: Consecutive adult ICU patients with delirium according to the CAM-ICU.

Intervention: Increasing dosage of rivastigmine or placebo as add-on medication.

Primary study parameters: Duration of delirium. Secondary study parameters: Delirium severity, length of ICU and hospital stay, functional status and mortality after 3 months.

Sample size: 440 patients will be included. Economic evaluation: includes a comparison of direct and indirect medical costs.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Burden: questionnaires (duration: 30 minutes). Risk: possible exposure to drug not indicated for the disorder. Benefit: possible treatment with according to experts possible beneficial drug. Consideration: The investigators of this study believe that the burden and risk do not exceed the expected benefit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Positive CAM-ICU

Exclusion Criteria:

* Known allergy to rivastigmine
* Unable to receive enteric medication
* Pregnant or lactating
* Renal replacement therapy
* Hepatic encephalopathy
* Second or third degree atrioventricular block
* Uncertainty about diagnosis delirium and no confirmation by neurologist, psychiatrist or geriatrician
* Parkinson's disease.
* Lewy body dementia.
* ECG QT interval above 500 msec.
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Duration of delirium | 3 months

SECONDARY OUTCOMES:
Severity of delirium | 3 months
Use of physical restraints | 3 months
Use of escape medication (i.c. Haloperidol or benzodiazepines) | 3 months
Number of accidental removed catheters | 3 months
Length of ICU stay | 3 months
Length of in-hospital stay | 3 months
Cognitive outcomes | 3 months
Activity of daily living | 3 months
Healthcare costs | 3 months
Frequency and distribution of side effects | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Arjen JC Slooter, MD. PhD., Principal Investigator — University Medical Center Utrecht, the Netherlands
Locations (6):
- Netherlands (6):
  - Gelre Hospitals; lukas site, Apeldoorn, Gelderland
  - Medical Center Alkmaar, Alkmaar, North Holland
  - Medical Center Leeuwarden, Leeuwarden, Provincie Friesland
  - Erasmus Medical Center, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht
  - Diakonessenhuis, Utrecht, Utrecht

REFERENCES:
- [Derived] van Eijk MM, Roes KC, Honing ML, Kuiper MA, Karakus A, van der Jagt M, Spronk PE, van Gool WA, van der Mast RC, Kesecioglu J, Slooter AJ. Effect of rivastigmine as an adjunct to usual care with haloperidol on duration of delirium and mortality in critically ill patients: a multicentre, double-blind, placebo-controlled randomised trial. Lancet. 2010 Nov 27;376(9755):1829-37. doi: 10.1016/S0140-6736(10)61855-7. Epub 2010 Nov 4. PMID 21056464